CLINICAL TRIAL: NCT00111761
Title: A Clinical Trial of the Safety and Efficacy of ABX-EGF in Combination With Irinotecan, Leucovorin, and 5-Fluorouracil in Subjects With Metastatic Colorectal Cancer
Brief Title: Evaluating Panitumumab (ABX-EGF) in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20025409; NCT00047151 (obsolete NCT alias)
Record Dates: First submitted 2005-05-25; First posted 2005-05-26 (Estimated); Results first posted 2011-06-03 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-11

CONDITIONS: Colorectal Cancer
Keywords: Immunex; Panitumumab; ABX-EGF; Abgenix
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Panitumumab; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1: Panitumumab + IFL (Experimental): Panitumumab (2.5 mg/kg once weekly for up to 48 weeks or until disease progression, intolerable adverse event or other reason for discontinuation) in combination with irinotecan, 5-fluorouracil (5-FU)and leucovorin (IFL chemotherapy regimen)
  Interventions: Drug: Irinotecan; Biological: Panitumumab; Drug: 5-Fluorouracil; Drug: Leucovorin
- Part 2: Panitumumab + FOLFIRI (Experimental): Panitumumab (2.5 mg/kg once weekly until disease progression, intolerable adverse event or other reason for discontinuation) in combination with irinotecan/5-FU/leucovorin chemotherapy (the FOLFIRI regimen)
  Interventions: Drug: Irinotecan; Biological: Panitumumab; Drug: 5-Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Irinotecan — Part 1: 125 mg/m^2 IV infusion once a week on weeks 1 through 4 of each 6-week treatment cycle. Part 2: 180 mg/m^2 IV infusion every other week until disease progression or unable to tolerate.
Biological: Panitumumab — Intravenous (IV) infusions of panitumumab 2.5 mg/kg once a week delivered in 6-week cycles.
  Other Names: ABX-EGF
Drug: 5-Fluorouracil — Part 1: IV bolus 500 mg/m^2 on weeks 1 through 4 of each 6-week cycle. Part 2: IV bolus 400 mg/m^2 and infusional 2400-3000 mg/m^2 over 46 hours once every other week until disease progression or unable to tolerate.
Drug: Leucovorin — Part 1: IV bolus 20 mg/m^2 on weeks 1 through 4 of each 6-week cycle. Part 2: 400 mg/m^2 every other week until disease progression or unable to tolerate.

SUMMARY:
The purpose of this study is to determine if panitumumab, in combination with irinotecan, leucovorin, and 5-fluorouracil (5-FU) is safe and efficacious in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Indication Metastatic Colorectal Cancer Primary Objective To assess the safety of ABX-EGF in combination with the FOLFIRI regimen in subjects with metastatic colorectal cancer. (The primary objective in the original protocol was to assess progression free survival after treatment with ABX-EGF in combination with the Saltz regimen in subjects with metastatic colorectal cancer).

Secondary Objective(s) To assess the clinical efficacy of ABX-EGF in combination with the FOLFIRI regimen in subjects with metastatic colorectal cancer. (Secondary objectives in the original protocol were to assess safety and additional measures of the clinical efficacy of ABX-EGF in combination with the Saltz regimen in subjects with metastatic colorectal cancer).

To assess the pharmacokinetics (PK) of ABX-EGF in combination with the FOLFIRI regimen in subjects with metastatic colorectal cancer. (Secondary objectives in the original protocol were to assess the PK of ABX-EGF in combination with the Saltz regimen, and the PK of irinotecan (IR) and its active metabolite SN-38 when IR is given in combination with ABX-EGF, leucovorin (LV), and 5-fluorouracil (5-FU) in subjects with metastatic colorectal cancer)

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and sign an Institutional Review Board (IRB)-approved informed consent form
* Pathologic diagnosis of colorectal cancer - Metastatic colorectal adenocarcinoma
* If history of adjuvant chemotherapy for colorectal cancer, must have been free of disease for greater than or equal to 1 year after completion of adjuvant chemotherapy
* Unidimensionally measurable disease
* Paraffin-embedded tumor tissue available for immunohistochemistry studies of epidermal growth factor receptor (EGFr) expression (archived tissue is acceptable)
* Tumor over-expressing EGFr by immunohistochemistry (staining must be the sum of 1+, 2+ and 3+ in greater than or equal to 10% of evaluated tumor cells; staining and evaluation to be conducted at a central laboratory)
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1
* Adequate hematologic, renal, and hepatic function

Exclusion Criteria:

* Female (of childbearing potential, post-menopausal for less than 6 months, not surgically sterilized, or not abstinent) not consenting to use adequate contraceptive precautions during the course of the study and for 6 months after the last ABX-EGF infusion
* Female who is breast-feeding or pregnant
* Any kind of disorder that compromises the ability of the patient to give written informed consent and/or comply with the study procedures
* History of any chronic medical or psychiatric condition or laboratory abnormality that, in the opinion of the investigator, may increase the risks associated with study participation or study drug administration or may interfere with compliance or the interpretation of study results
* Untreated brain metastases
* Therapy for colorectal cancer other than surgery and 5-FU-based adjuvant therapy
* Prior treatment for metastatic colorectal cancer
* Prior irinotecan
* Prior or concurrent radiation therapy for colorectal cancer, including prior adjuvant radiation therapy to the pelvis
* Known allergy to irinotecan, 5-fluorouracil, or leucovorin
* Known Gilbert's disease
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Prior EGFr-targeting agents
* Use of investigational therapy used with adjuvant intent within 30 days before the first ABX-EGF infusion
* If prior history of cancer other than colorectal carcinoma, basal cell carcinoma, or cervical carcinoma in situ, no treatment or active disease within 5 years
* Active inflammatory bowel disease or other bowel disease (other than colorectal carcinoma) causing chronic diarrhea (defined as greater than 4 stools per day)
* Partial or complete bowel obstruction, known chronic malabsorption, total colectomy, or other major abdominal surgery that might result in substantial alteration in transit to absorption of oral medication
* Ascites or pleural effusion requiring therapeutic paracentesis or thoracentesis; subject with small, stable, asymptomatic pleural effusions or ascites may be enrolled; subject who has been rendered asymptomatic by successful sclerosis of an effusion may be enrolled.
* Active interstitial pneumonia or interstitial fibrosis
* Left ventricular ejection fraction (LVEF) less than 45%, as measured by multiple-gated acquisition (MUGA) scan - Myocardial infarction within 1 year before the first ABX-EGF infusion
* Any of the following within 6 months before the first study drug dose:

  * Unstable angina;
  * Symptomatic congestive heart failure;
  * Serious uncontrolled cardiac arrhythmia;
  * Cerebrovascular accident or transient ischemic attack;
  * Pulmonary embolism;
  * Deep vein thrombosis;
  * Other significant thromboembolic event.
* Subject known to be human immunodeficiency virus (HIV) positive
* History of any chronic medical or psychiatric condition or laboratory abnormality that, in the opinion of the Investigator, may increase the risks associated with study participation or study drug administration or may interfere with patient compliance or the interpretation of study results
* Unwilling or unable to comply with study requirements
* Known allergy to the ingredients of the study drug or to Staphylococcus protein A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2002-07; Primary Completion 2008-02 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Berlin J, Posey J, Tchekmedyian S, Hu E, Chan D, Malik I, Yang L, Amado RG, Hecht JR. Panitumumab with irinotecan/leucovorin/5-fluorouracil for first-line treatment of metastatic colorectal cancer. Clin Colorectal Cancer. 2007 Mar;6(6):427-32. doi: 10.3816/CCC.2007.n.011. PMID 17531105
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: FDA-approved Drug Labeling — http://www.vectibix.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 19 Jul 2002 through 20 April 2004
Groups:
- Panitumumab With FOLFIRI: Panitumumab (2.5 mg/kg once weekly until disease progression, intolerable adverse event or other reason for discontinuation) in combination with irinotecan/5-FU/leucovorin chemotherapy (the FOLFIRI regimen)
- Panitumumab With IFL: Panitumumab (2.5 mg/kg once weekly for up to 48 weeks or until disease progression, intolerable adverse event or other reason for discontinuation) in combination with irinotecan, 5-fluorouracil and leucovorin (IFL chemotherapy regimen)
Period: Part 1
Arm/Group | Panitumumab With FOLFIRI | Panitumumab With IFL
Started | 0 (This treatment group was not initiated until Part 2) | 19
Completed | 0 | 14 (Completed through safety followup)
Not Completed | 0 | 5
Not completed — Physician Decision | 0 | 1
Not completed — Death | 0 | 2
Not completed — Other | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Part 2
Arm/Group | Panitumumab With FOLFIRI | Panitumumab With IFL
Started | 24 | 0 (This treatment group was used in Part 1 only)
Completed | 16 | 0
Not Completed | 8 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 0
Not completed — Disease progression | 3 | 0
Not completed — Protocol-specified criteria | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Panitumumab With IFL: Panitumumab in combination with irinotecan, 5-fluorouracil and leucovorin (IFL chemotherapy regimen)
- Panitumumab With FOLFIRI: Panitumumab in combination with irinotecan/5-FU/leucovorin chemotherapy (the FOLFIRI regimen)
- Total: Total of all reporting groups
Arm/Group | Panitumumab With IFL | Panitumumab With FOLFIRI | Total
Number analyzed (Participants) | 19 | 24 | 43
Age Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (12.1) | 60.7 (15.0) | 58.9 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 16 | 14 | 30
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 1 | 2
  Black or African American | 4 | 3 | 7
  Hispanic or Latino | 1 | 2 | 3
  White or Caucasian | 13 | 18 | 31
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 or Grade 4 Diarrhea (Part 2)
Description: The number of participants with grade 3 or grade 4 diarrhea in Part 2 of the study. Grading of diarrhea followed the grading scale in Version 2.0 of the National Cancer Institute Common Toxicity Criteria (NCI CTC).
Time Frame: Until disease progression (median 47 weeks)
Population: Subjects Treated Analysis Set, composed of participants who received at least one dose of panitumumab or one dose of chemotherapy.
Measure: Number; unit: Participants
Arm/Group | Panitumumab With FOLFIRI
Number analyzed (Participants) | 24
Participants | 6
Statistical Analysis 1: Comparison: Panitumumab With FOLFIRI; Test type: Superiority or Other; Percentage of participants = 25.0, 95% CI [9.8 to 46.7]

2. Primary Outcome: Number of Participants With Grade 3 or Grade 4 Diarrhea (Part 1)
Description: The number of participants with grade 3 or grade 4 diarrhea in Part 1 of the study. Grading of diarrhea followed the grading scale in Version 2.0 of the National Cancer Institute Common Toxicity Criteria (NCI CTC).
Time Frame: Until disease progression (median 35 weeks) or 48 weeks, whichever occurred first
Population: Subjects Treated Analysis Set, composed of all consented participants who received at least 1 dose of panitumumab and at least 1 dose of chemotherapy.
Measure: Number; unit: Participants
Arm/Group | Panitumumab With IFL
Number analyzed (Participants) | 19
Participants | 11
Statistical Analysis 1: Comparison: Panitumumab With IFL; Test type: Superiority or Other; Percentage of participants = 58, 95% CI [34 to 80]

3. Secondary Outcome: Number of Participants With an Objective Tumor Response (Part 2)
Description: Objective tumor response (complete or partial) in Part 2 of the study, based on Response Evaluation Criteria in Solid Tumors (RECIST), where complete response = disappearance of all target lesions, partial response = ≥30% reduction in lesion size, progressive disease = ≥20% increase in tumor size; otherwise stable disease.
Time Frame: Until disease progression (median 47 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Panitumumab With FOLFIRI
Number analyzed (Participants) | 24
Participants | 8
Statistical Analysis 1: Comparison: Panitumumab With FOLFIRI; Test type: Superiority or Other; Percentage = 33.3, 95% CI [15.6 to 55.3]

4. Secondary Outcome: Time to Disease Progression (Part 2)
Description: Kaplan-Meier estimate of median time from the first dose of study drug to first observed disease progression or death if the death was due to disease progression (whichever comes first) in Part 2 of the study. Participants who had not progressed or died for reasons other than disease progression were censored at their last disease assessment date.
Time Frame: From enrollment until death or diease progression. Maximum follow-up time was 16 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab With FOLFIRI
Number analyzed (Participants) | 24
weeks | 47.3 [26.0 to NA] — Could not be estimated due to the low number of events.

5. Secondary Outcome: Progression-free Survival Time (Part 2)
Description: Kaplan-Meier estimate of median time from enrollment to death or disease progression in Part 2 of the study. Participants who had not progressed and had not died were censored at their last disease assessment date.
Time Frame: From enrollment until disease progression or death. Maximum follow-up time was 16 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab With FOLFIRI
Number analyzed (Participants) | 24
weeks | 41.1 [26.0 to NA] — Could not be estimated due to the low number of events.

6. Secondary Outcome: Survival Time (Part 2)
Description: Kaplan-Meier estimate of the median time from enrollment to death from any cause. Participants who did not die on study were censored at their last contact date.
Time Frame: From enrollment until death. Maximum follow-up time was 16 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab With IFL
Number analyzed (Participants) | 19
weeks | 73.1 [59.4 to NA] — Could not be estimated due to the low number of events.

7. Secondary Outcome: Number of Participants Who Died (Part 2)
Description: The number of participants in Part 2 who died during the study.
Time Frame: From enrollment until last contact. Maximum follow-up was 16 months.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Panitumumab With FOLFIRI
Number analyzed (Participants) | 24
participants | 6

8. Secondary Outcome: Number of Participants With Objective Tumor Response (Part 1)
Description: Objective tumor response (complete or partial) in Part 1 of the study, based on Response Evaluation Criteria in Solid Tumors (RECIST), where complete response = disappearance of all target lesions, partial response = ≥30% reduction in lesion size, progressive disease = ≥20% increase in tumor size; otherwise stable disease.
Time Frame: Until disease progression (median 35 weeks) or 48 weeks, whichever occurred first
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Panitumumab With IFL
Number analyzed (Participants) | 19
Participants | 9
Statistical Analysis 1: Comparison: Panitumumab With IFL; Test type: Superiority or Other; Percentage of participants = 47.4, 95% CI [24.4 to 71.1]

9. Secondary Outcome: Progression-free Survival Time (Part 1)
Description: Kaplan-Meier estimate of median time from enrollment to death or disease progression in Part 1 of the study. Participants who had not progressed and had not died were censored at their last disease assessment date.
Time Frame: From enrollment until disease progression or death. Maximum follow-up time was 25 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab With IFL
Number analyzed (Participants) | 19
weeks | 24.3 [19.0 to 36.0]

10. Secondary Outcome: Time to Disease Progression (Part 1)
Description: Kaplan-Meier estimate of the median time from the first dose of study drug to disease progression or death if due to disease progression (whichever comes first) in Part 1 of the study. Participants who had not progressed or died for reasons other than disease progression were censored at their last disease assessment date.
Time Frame: From enrollment until disease progression or death. Maximum follow-up time was 25 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab With IFL
Number analyzed (Participants) | 19
weeks | 35.0 [21.7 to 72.0]

11. Secondary Outcome: Survival Time (Part 1)
Description: as for outcome 6
Time Frame: From enrollment until death. Maximum follow-up time was 25 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab With IFL
Number analyzed (Participants) | 19
weeks | 73.1 [59.4 to NA] — Could not be estimated due to the low number of events.

12. Secondary Outcome: Time to Treatment Failure (Part 1)
Description: Kaplan-Meier estimate of the median time from the date of first dose of panitumumab or chemotherapy to the date the decision was made to end treatment for any reason in Part 1 of the study.
Time Frame: Until disease progression (median 35 weeks) or 48 weeks, whichever occurred first
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Panitumumab With IFL
Number analyzed (Participants) | 19
Weeks | 24.3 [7.9 to 36.0]

13. Secondary Outcome: Time to Initial Objective Tumor Response (Part 1)
Description: Median time to first observed objective tumor response (complete or partial) among responders in Part 1 of the study.
Time Frame: Until disease progression (median 35 weeks) or 48 weeks, whichever occurred first
Population: Subset of Subjects Treated Analysis Set, composed of all consented participants who received at least 1 dose of panitumumab and at least 1 dose of chemotherapy, who had an objective tumor response.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Panitumumab With IFL
Number analyzed (Participants) | 9
weeks | 5.9 [5.4 to 11.3]

ADVERSE EVENTS:
Time Frame: First dose through maximum of safety FU or 30 days after last dose (median 47 weeks follow-up)
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Panitumumab Plus IFL | Panitumumab Plus FOLFIRI
Serious Adverse Events (participants affected / at risk) | 12/19 | 11/24
Other Adverse Events (participants affected / at risk) | 19/19 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus IFL (N=19) | Panitumumab Plus FOLFIRI (N=24)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Coagulation time prolonged (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus IFL (N=19) | Panitumumab Plus FOLFIRI (N=24)
Anaemia (Blood and lymphatic system disorders) | 6 | 3
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 6 | 3
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Palpitations (Cardiac disorders) | 1 | 1
Blepharitis (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 4
Diplopia (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 2 | 0
Eye pruritus (Eye disorders) | 0 | 3
Eyelid oedema (Eye disorders) | 0 | 2
Growth of eyelashes (Eye disorders) | 1 | 0
Keratoconjunctivitis sicca (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 2
Vision blurred (Eye disorders) | 2 | 4
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 8
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Anal discomfort (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 7 | 10
Defaecation urgency (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 16 | 19
Dry mouth (Gastrointestinal disorders) | 1 | 6
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Dysphagia (Gastrointestinal disorders) | 2 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 4 | 4
Frequent bowel movements (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Glossodynia (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 3 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 2
Hypertrophy of tongue papillae (Gastrointestinal disorders) | 1 | 0
Intestinal stenosis (Gastrointestinal disorders) | 1 | 0
Loose stools (Gastrointestinal disorders) | 3 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 13 | 15
Oral pain (Gastrointestinal disorders) | 2 | 4
Proctalgia (Gastrointestinal disorders) | 1 | 1
Rectal discharge (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 5 | 1
Retching (Gastrointestinal disorders) | 0 | 2
Sensitivity of teeth (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 8 | 6
Vomiting (Gastrointestinal disorders) | 5 | 11
Asthenia (General disorders) | 2 | 6
Catheter site pain (General disorders) | 0 | 2
Chest discomfort (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 2
Fatigue (General disorders) | 16 | 19
Influenza like illness (General disorders) | 1 | 0
Infusion site pain (General disorders) | 1 | 0
Infusion site reaction (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 9
Oedema (General disorders) | 0 | 3
Oedema peripheral (General disorders) | 7 | 4
Pain (General disorders) | 3 | 3
Pyrexia (General disorders) | 5 | 5
Rigors (General disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 2
Cellulitis orbital (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 1
Fungal infection (Infections and infestations) | 1 | 1
Fungal skin infection (Infections and infestations) | 0 | 2
Furuncle (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Genital candidiasis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 2 | 2
Nail infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1
Paronychia (Infections and infestations) | 4 | 1
Pharyngitis (Infections and infestations) | 2 | 0
Rash pustular (Infections and infestations) | 0 | 4
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 0 | 5
Skin laceration (Injury, poisoning and procedural complications) | 0 | 3
Alanine aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Ejection fraction abnormal (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 3 | 4
Anorexia (Metabolism and nutrition disorders) | 7 | 13
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 4 | 5
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Facial pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Local swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Ageusia (Nervous system disorders) | 1 | 0
Cholinergic syndrome (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 6 | 8
Dysgeusia (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 2 | 5
Hypoaesthesia (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 3
Syncope (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 3
Depression (Psychiatric disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 2 | 7
Mood swings (Psychiatric disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 3
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 10
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 10
Erythema (Skin and subcutaneous tissue disorders) | 1 | 6
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 2
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 9
Rash (Skin and subcutaneous tissue disorders) | 16 | 19
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 5 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 4
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 6
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2
Hot flush (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 3 | 3
Phlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.